CLINICAL TRIAL: NCT00158769
Title: An Open-Label, Non-Randomised, Pharmacokinetic, Metabolic Disposition and Safety Study of a 3 Day Continuous Infusion of GR270773 in Healthy Subjects and Subjects With Hepatic Impairment.
Brief Title: A Study To Compare The Effects Of The Infusion Of A Sepsis Drug Between Healthy Adults And Adults With Damaged Livers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD10007
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Sepsis
Keywords: Hepatic Impairment; GR270773; Emulsion
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects with moderate hepatic impairment (Experimental): Subjects with moderate hepatic impairment as defined by a Child-Pugh score of 7-9 will be included. Subjects will be given GR270773 as a loading infusion of 25 milligram per kilogram per hour (mg/kg/hr) for 2 hours followed by a maintenance infusion of 5 mg/kg/hr for 70 hours.
  Interventions: Drug: Intravenous GR270773 - Phospholipid emulsion
- Healthy subjects (Experimental): Subjects will be matched as closely as possible to the group of moderate hepatic subjects for gender, age and body mass index (BMI). Subjects will be administered 25 mg/kg/hr GR270773 as a loading dose for 2 hours followed by a maintenance infusion of 5 mg/kg/hr for 70 hours. Following a washout period of 21 days, the subjects will then receive a loading dose of 75 mg/kg/hr for 2 hours followed by a maintenance dose of 12.5 mg/kg/hr of GR270773 for 70 hours.
  Interventions: Drug: Intravenous GR270773 - Phospholipid emulsion

INTERVENTIONS:
Drug: Intravenous GR270773 - Phospholipid emulsion — GR270773 (lipid emulsion) is a sterile, white to off-white, semi-translucent liquid for intravenous injection.

SUMMARY:
This compound, GR270773, is a lipid based compound being developed to treat Sepsis. Lipids are broken down in the body by the liver. This study is designed to see whether the effect of the drug in people with poorly functioning livers is any different to the effect on healthy adults.

ELIGIBILITY:
Inclusion criteria:

* Patients with known history of liver disease (either with or without history of alcohol abuse).
* Previous confirmation of liver cirrhosis by liver biopsy or other medical imaging technique.
* Child-Pugh score of 7-9 (moderate impairment) BMI 19-29 Kg/m2.
* Healthy volunteers to match the hepatically impaired subjects in a 1:1 ratio by gender, age, BMI.

Exclusion criteria:

* Lactating or pregnant females.
* Subjects with BP > 160/90.
* Subjects who, within the past six months, have had a history of significant drug or alcohol abuse, or any indication of regular use of more than 14 units of alcohol per week for women, or 21 units/week for men.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2005-03-31 (Actual); Primary Completion 2005-10-26 (Actual); Study Completion 2005-10-26 (Actual)

PRIMARY OUTCOMES:
Compare drug concentrations in the blood between patients with impaired liver function and normal healthy adults, after 72 hours. Determine whether administration of study drug alters the lipid make-up of healthy adults in any way. | Up to Day 16

SECONDARY OUTCOMES:
Determine drug concentrations in blood after 2 hour run-in period and after 72 hour infusion period. Determine whether administration of study drug alters the lipid make-up of patients with impaired liver function in any way. | Up to Day 16

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bratislava, Slovakia

REFERENCES:
- See also: Results for study EMD10007 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/EMD10007?search=study&search_terms=EMD10007#rs